CLINICAL TRIAL: NCT02346617
Title: Adoptive Transfer of pp65-specific T Cells for the Treatment of Refractory Cytomegalovirus (CMV) Infection in Allogeneic Hematopoietic Cell Transplant Recipients
Brief Title: Adoptive Transfer of pp65-specific T Cells for the Treatment of Refractory Cytomegalovirus (CMV) Infection
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the KoreaFDA issue
Sponsor: Yae-Jean Kim (Other)
Collaborators: Miltenyi Biotec B.V. & Co. KG (Industry)
Responsible Party: Sponsor-Investigator, Yae-Jean Kim, Associate professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2010-08-129-008
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Cytomegalovirus Infections
Keywords: CMV; T cell therapy
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allogeneic HSCT (Experimental): The present study will investigate in a single-center (Samsung Medical Center), open-label, single arm by direct infusions of donor-derived CMV-spefic IFN-γ positive T-cells for the treatment of refractory CMV infection in allogeneic hematopoietic stem cell transplant (HSCT) recipients.
  Interventions: Biological: IFN-γ positive selected T-cells

INTERVENTIONS:
Biological: IFN-γ positive selected T-cells — No intervention

SUMMARY:
To evaluate the safety and efficacy for treatment of persistent CMV infection in hematopoietic cell transplant (HCT) recipients.

DETAILED DESCRIPTION:
HCT recipients who are receiving immunosuppressive agents to control graft versus host diseases (GVHD) are at high risk for serious CMV infection due to CMV reactivation or reinfection during their post-transplant period.

Antiviral agents used to treat CMV infection have well-known side effects such as bone marrow suppression causing cytopenia and renal toxicities. Therefore, patients in a serious condition would have a higher probability of antiviral treatment-related toxicities and also increased possibility for prolonged antiviral treatment, thus development of antiviral resistance and risk of treatment failure.

Allogeneic HCT recipients are typically lack of these CMV-specific T cells during the post-transplant period and their immune function can be further repressed especially when they are on additional immunosuppressive agents to prevent GVHD. Therefore, these patients may benefit from CMV-specific T cell adoptive transfer.

ELIGIBILITY:
Inclusion Criteria:

* Less than 66 years old Allogeneic HCT recipients who received stem cells from related CMV positive serology donors
* AND recipients have persistent CMV infection more than 2 weeks on antiviral treatment

Exclusion Criteria:

* HCT recipients with severe graft versus host disease, grade 3 or more
* OR organ dysfunction (brain, heart, lung, liver, and kidney): altered mentality, extracorporeal membrane oxygenation, mechanical ventilator, increased liver enzymes 5 times above upper normal values, bilirubin level >3 mg/dL, CrCl < 30 mL/min

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Level of enriched IFN-Υ+ T-cells upon pp65 stimulation | 2 weeks

SECONDARY OUTCOMES:
Treatment efficacy of CMV infection, defined as reduction of CMV viremia, ex vivo enrichment of CMV antigen (pp65) -specific T cells in peripheral blood. | 2 weeks
  Treatment efficacy defined as reduction of CMV viremia, ex vivo enrichment of CMV antigen (pp65) -specific T cells in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Yae-Jean Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-Gu, South Korea

REFERENCES:
- [Background] Kim YJ, Boeckh M, Cook L, Stempel H, Jerome KR, Boucek R Jr, Burroughs L, Englund JA. Cytomegalovirus infection and ganciclovir resistance caused by UL97 mutations in pediatric transplant recipients. Transpl Infect Dis. 2012 Dec;14(6):611-7. doi: 10.1111/j.1399-3062.2012.00760.x. PMID 23198963
- [Background] Feuchtinger T, Opherk K, Bethge WA, Topp MS, Schuster FR, Weissinger EM, Mohty M, Or R, Maschan M, Schumm M, Hamprecht K, Handgretinger R, Lang P, Einsele H. Adoptive transfer of pp65-specific T cells for the treatment of chemorefractory cytomegalovirus disease or reactivation after haploidentical and matched unrelated stem cell transplantation. Blood. 2010 Nov 18;116(20):4360-7. doi: 10.1182/blood-2010-01-262089. Epub 2010 Jul 12. PMID 20625005
- [Background] Peggs KS, Thomson K, Samuel E, Dyer G, Armoogum J, Chakraverty R, Pang K, Mackinnon S, Lowdell MW. Directly selected cytomegalovirus-reactive donor T cells confer rapid and safe systemic reconstitution of virus-specific immunity following stem cell transplantation. Clin Infect Dis. 2011 Jan 1;52(1):49-57. doi: 10.1093/cid/ciq042. PMID 21148519
- [Background] Peggs KS, Verfuerth S, Pizzey A, Chow SL, Thomson K, Mackinnon S. Cytomegalovirus-specific T cell immunotherapy promotes restoration of durable functional antiviral immunity following allogeneic stem cell transplantation. Clin Infect Dis. 2009 Dec 15;49(12):1851-60. doi: 10.1086/648422. PMID 19911966
- [Background] Yi ES, Kim YJ. Cytomegalovirus infection according to cell source after hematopoietic cell transplantation in pediatric patients. Yonsei Med J. 2012 Mar;53(2):393-400. doi: 10.3349/ymj.2012.53.2.393. PMID 22318829
- [Background] Tomblyn M, Chiller T, Einsele H, Gress R, Sepkowitz K, Storek J, Wingard JR, Young JA, Boeckh MJ; Center for International Blood and Marrow Research; National Marrow Donor program; European Blood and MarrowTransplant Group; American Society of Blood and Marrow Transplantation; Canadian Blood and Marrow Transplant Group; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America; Association of Medical Microbiology and Infectious Disease Canada; Centers for Disease Control and Prevention. Guidelines for preventing infectious complications among hematopoietic cell transplantation recipients: a global perspective. Biol Blood Marrow Transplant. 2009 Oct;15(10):1143-238. doi: 10.1016/j.bbmt.2009.06.019. No abstract available. PMID 19747629
- [Background] Boeckh M, Ljungman P. How we treat cytomegalovirus in hematopoietic cell transplant recipients. Blood. 2009 Jun 4;113(23):5711-9. doi: 10.1182/blood-2008-10-143560. Epub 2009 Mar 18. PMID 19299333
- [Background] Vivier E, Ugolini S. Natural killer cells: from basic research to treatments. Front Immunol. 2011 Jun 3;2:18. doi: 10.3389/fimmu.2011.00018. eCollection 2011. No abstract available. PMID 22566808
- [Background] Hadaya K, Avila Y, Valloton L, de Rham C, Bandelier C, Ferrari-Lacraz S, Pascual M, Pantaleo G, Martin PY, Buhler L, Villard J. Natural killer cell receptor--repertoire and functions after induction therapy by polyclonal rabbit anti-thymocyte globulin in unsensitized kidney transplant recipients. Clin Immunol. 2010 Nov;137(2):250-60. doi: 10.1016/j.clim.2010.07.004. Epub 2010 Aug 17. PMID 20719569
- [Background] Vacher-Coponat H, Brunet C, Moal V, Loundou A, Bonnet E, Lyonnet L, Ravet S, Sampol-Manos E, Sampol J, Berland Y, George FD, Paul P. Tacrolimus/mycophenolate mofetil improved natural killer lymphocyte reconstitution one year after kidney transplant by reference to cyclosporine/azathioprine. Transplantation. 2006 Aug 27;82(4):558-66. doi: 10.1097/01.tp.0000229390.01369.4a. PMID 16926601